CLINICAL TRIAL: NCT03953573
Title: Management of Post-delivery Pain and Its Impact on Resumption of Sexuality
Acronym: SMD
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_0057
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Sexuality; Delivery
MeSH Terms: conditions — Sexuality | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women post-delivery
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey completed at 1 day, 8 days 1 or 3 months post delivery

SUMMARY:
Study of management of pain and information given to women post-delivery and their impact of the resumption of sexuality.

Survey to be completed by women at 8 and 15 days and 1 or 3 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous woman
* Age between 18 and 45 years old
* Delivery after 37 weeks of amenorrhea
* Speaking French
* Pregnancy, delivery and new-born examination without morphologic or biometric abnormalities, respiratory distress and no pathology discovered at neonatal screening on day 3
* Heterosexual woman with partner
* Signed consent
* Affiliate of national health insurance scheme

Exclusion Criteria:

* Multiple pregnancy,
* BMI > 30
* Conjugopathie
* Known psychiatric history
* Medical history with gynecologic impact
* Surgery history with gynecologic impacts
* Hysterectomy post-delivery
* Protected by French law

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primiparous women, delivery at hospital.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Post-delivery sexuality resumption | 3 months
  Time to sexuality resumption

SECONDARY OUTCOMES:
Discussion with healthcare professional on post-delivery sexuality | 1 month
  Number of women receiving advice from a health professional
Pain post-delivery | 3 months
  Number of women needed pain treatment or with problem for sexuality resumption
Sexual health | 3 months
  Frequency of sex

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No